CLINICAL TRIAL: NCT05261568
Title: The Effect of Progressive Relaxation Exercises on Fatigue and Sleep Quality in Individuals With Epilepsy
Brief Title: The Effect of Progressive Relaxation Exercises on Fatigue and Sleep Quality in İndividuals With Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Neşe İŞCAN AYYILDIZ, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Supportive Care
Other Study IDs: AtaturkUnıversıty Nusing
Record Dates: First submitted 2022-01-14; First posted 2022-03-02 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Epilepsy; Sleep; Fatigue
MeSH Terms: conditions — Epilepsy; Fatigue

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The first application is carried out by a researcher close to the polyclinic with care and demonstration.
  The application will be suggested by hanging it from side to side in sitting position. They will be informed about the same application conditions in their own practice at home.
  The program, which will last for 6 weeks, will continue from the home environment after a video surveillance observed by the beneficiary.
  Periods of entry and exit times thanks to the mobile program. It will be done over the phone by the people who will come for 6 weeks. history book, lack of tools, etc. a website will be searched. Adhering to application products through study. A total of 42 sessions for 6 weeks, 7 days a week. About 30min. It is used to benefit from training to benefit from sustained progression. Apart from that, he can enjoy wearing it by dressing casually and casually.
  Interventions: Behavioral: PROGRESSIVE RELAXATION EXERCISE
- control gruop (No Intervention): The control group did not receive any intervention other than their own treatment during the study.
  will not be applied. Progressive relaxation exercise application to the individuals included in the control group personal information form, Pittsburgh sleep quality index, fatigue severity scale will be applied as test-post-test.

INTERVENTIONS:
Behavioral: PROGRESSIVE RELAXATION EXERCISE — Progressive relaxation exercise will be done for 6 weeks by watching the animation video in the mobile application program.
  Arms: experimental group

SUMMARY:
Aim: It was conducted to determine the effect of web-based animation supported progressive relaxation exercise on fatigue and sleep quality in individuals with epilepsy. Material and Methods: As a randomized controlled study with a pretest- posttest model, it was conducted with individuals with epilepsy who applied to Giresun University Faculty of Medicine Neurology Outpatient Clinic between February and December 2022.The sample of the study was determined as 60 epilepsy patients, 30 of which were in the control-30 experimental group, using power analysis. The data were collected by face-to-face interview technique using Personal Information Form, Pittsburg Sleep Quality Index, Fatigue Severity Scale.

ELIGIBILITY:
Inclusion Criteria:

* be over the age of 18
* Having been diagnosed with epilepsy for at least 6 months
* Individuals with an average score of 4.1 or higher on the fatigue severity scale
* Individuals with a Pittsburg Sleep Quality Index total score above 5
* Being able to use mobile phone (IOS-Android)
* Being able to speak Turkish
* Up to 6 months before the study, techniques such as meditation, hypnosis, yoga not benefited,
* Having a neurological, systemic and psychiatric disease other than epilepsy not to be.

Exclusion Criteria:

* Not using a mobile phone,
* Up to 6 months before the study, techniques such as meditation, hypnosis, yoga to have benefited,
* Having a neurological, systemic and psychiatric disease other than epilepsy be.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
fatigue severity scale | An average of 1 year
  finished

SECONDARY OUTCOMES:
pittsburg sleep quality scale | An average of 1 year
  finished

CONTACTS AND LOCATIONS:
Overall Officials: Nuray DAYAPOĞLU, Principal Investigator — Ataturk University
Locations (1):
- Giresun Training and Research Hospital, Giresun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No